CLINICAL TRIAL: NCT02279147
Title: The Prevention and Treatment of SIRS in Patients With Cholestatic Jaundice After Operation.
Brief Title: Cholinergic Anti-inflammatory Pathway in Prevention & Treatment of the SIRS in Patients With Jaundice After Operation.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wanqing Gu (Other)
Responsible Party: Sponsor-Investigator, Wanqing Gu, The Prevention and Treatment of SIRS in Patients With Cholestatic Jaundice After Operation., Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHN-PLAGH-WGu-001
Record Dates: First submitted 2014-09-22; First posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Systemic Inflammatory Response Syndrome; Jaundice, Obstructive
Keywords: Systemic Inflammatory Response Syndrome; Jaundice, Obstructive; anti-inflammatory
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Jaundice, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- raceanisodamine & neostigmine (Experimental): Patients receive immediately raceanisodamine（10mg）by intramuscular injection after operation.Then the patients will be receive 50mg raceanisodamine and 0.15mg neostigmine within 24hs by slow injection into vein for three consecutive days.
  Interventions: Drug: neostigmine methylsulfate，raceanisodamine hydrochloride
- blank (No Intervention): Patients do not receive special treatment after operation.

INTERVENTIONS:
Drug: neostigmine methylsulfate，raceanisodamine hydrochloride — The patients receive immediately raceanisodamine hydrochloride(10mg) by intramuscular injection after operation .From that date, for three consecutive days, the patients will be receive 50mg raceanisodamine hydrochloride and 0.15mg neostigmine methylsulfate in the 24h by slow injection of vein.
  Arms: raceanisodamine & neostigmine

SUMMARY:
RATIONALE:Anticholinesterase drugs and cholinergic M receptor antagonist are applied to patients who have obstructive jaundice after operation.

PURPOSE:This clinical trial was designed to lower the incidence and mortality of operation complications in patients with obstructive jaundice .

DETAILED DESCRIPTION:
OBJECTIVES:

Ⅰ.Judge whether it has the effect of inhibiting inflammation, anti oxidative stress and anti apoptosis when the alpha 7 nicotinic acetylcholine receptors are activated .

Ⅱ.Judge whether it has the effect of reducing the incidence and mortality of operation complication when using Cholinesterase inhibitors and M cholinergic receptor blocking agent in Patients with obstructive jaundice after operation。

OUTLINE:Patients are assigned to 1 of 2 groups according to order of enrollment.

Group 1:Patients receive neostigmine methylsulfate and raceanisodamine hydrochloride on days 0,1,2 after operation.

Group 2:Patients do not receive any special treatment after operation.

All patients should be monitored the observed indexes on the day before the operation and one day, three days, five days after the operation.

ELIGIBILITY:
Inclusion Criteria:

Ⅰ.Accompanied by obstructive jaundice and plans to implement the liver resection of hilar bile duct carcinoma.

Patients with carcinoma of head of pancreas and plans to implement pancreaticoduodenectomy.

Ⅱ. Drugs which were used in the clinical trials is safe for patients.

Ⅲ.The patients did not occur the complication which would affect the experimental observation seriously after the operation.

Ⅳ.The patients agreed to participate in this clinical trial and sign the informed consent.

Exclusion Criteria:

Ⅰ.Patients are unwilling to accept the clinical trials or researchers believe that patients can not in compliance with the requirements of clinical research.

Ⅱ.Patients with tumor metastases widely or can not accept a predetermined operation scheme.

Ⅲ. The postoperative complications or other therapeutic measures take will affect the experimental observation seriously.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
C reactive protein | One year
  Indicator of the stress level.

SECONDARY OUTCOMES:
Temperature | One year
  Indicator of systemic inflammatory response syndrome.
Heart rate | One year
  Indicator of systemic inflammatory response syndrome.
Respiratory | One year
  Indicator of systemic inflammatory response syndrome.
PaCO2 | One year
  Indicator of systemic inflammatory response syndrome.
White blood cell count | one year
  Indicator of systemic inflammatory response syndrome.
Alanine aminotransferase（ALT) | One year
  Indicators of liver function.
Aspartate aminotransferase（AST） | One year
  Indicators of liver function.
Total bilirubin | One year
  Indicators of liver function.
Interleukin 1（IL-1） | One year
  Indicators of pro-inflammatory mediators
Interleukin 2（IL-2） | One year
  Pro-inflammatory mediators.
Interleukin 6（IL-6） | One year
  Pro-inflammatory mediators.
Interleukin 8（ IL-8） | One year
  Pro-inflammatory mediators
Tumor necrosis factor-α | One year
  Pro-inflammatory mediators.
Interleukin 10（ IL-10） | One year
  Anti-inflammatory mediators
Triiodothyronine(T3) & Thyroxin(T4) & Thyroid stimulating hormone(TSH) | One year
  Indicators of the stress level.

CONTACTS AND LOCATIONS:
Overall Officials: GU wanqing, Study Chair — CHN Chinese PLA General Hospital
Locations (1):
- CHN Chinese PLA General Hospital, Beijing, Beijing Municipality, China